CLINICAL TRIAL: NCT05496192
Title: A Phase II Study of Adjuvant Nivolumab Switch From Intravenous (IV) to Subcutaneous (SC) Use in Participants With Resected Stage III or Stage IV Melanoma or High Risk Invasive Urothelial Carcinoma Originating in the Bladder
Brief Title: A Study of Nivolumab Intravenous (IV) to Subcutaneous (SC) Switch in Adjuvant Melanoma and Bladder Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Replaced it with another clinical trial
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-6L6; 2022-000294-67 (EudraCT Number); U1111-1273-4725 (Registry Identifier: WHO)
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Melanoma; Urothelial Carcinoma
Keywords: Resected Invasive Urothelial Carcinoma; Nivolumab; Bladder; Melanoma; Adjuvant; Subcutaneous
MeSH Terms: conditions — Melanoma; Carcinoma, Transitional Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab IV followed by Nivolumab SC (Experimental)
  Interventions: Drug: Nivolumab/rHuPH20; Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab/rHuPH20 — Specified dose on specified days
  Other Names: Opdivo; BMS-986298
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558

SUMMARY:
The purpose of this study is to evaluate the switch from Nivolumab Intravenous (IV) infusions to Nivolumab Subcutaneous (SC) administration in participants with resected Stage IIIA/B/C/D or Stage IV melanoma or resected invasive Urothelial Carcinoma (UC) originating in the bladder who have high risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Participants must be eligible for adjuvant therapy for melanoma or muscle-invasive Urothelial Carcinoma (UC) originating from the bladder.
* All participants must have disease-free status (DFS) documented by a complete physical examination and imaging studies within 4 weeks prior to treatment assignment.

Exclusion Criteria:

* History of ocular or uveal or mucosal melanoma.
* Upper tract UC (ureter, renal pelvis), non-muscle-invasive UC.
* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to treatment assignment.
* Untreated/unresected Central Nervous System (CNS) or leptomeningeal metastases.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2024-06-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants That Prefer Nivolumab SC at the First Assessment of Patient Preference Using Patient Experience and Preference Questionnaire (PEPQ) (Question 1) | Up to 24 hours after first full dose at Cycle 4, Day 1 (98 Days)

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 100 days following last dose of nivolumab (Up to Day 465)
Proportion of Participants That Prefer Nivolumab SC at the Second Assessment of Patient Preference Using PEPQ (Question 1) | Up to 24 hours after fourth full dose at Cycle 5, Day 15 (140 Days)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Germany (2):
  - Local Institution - 0020, Essen, North Rhine-Westphalia
  - Local Institution - 0001, Berlin
- Local Institution - 0002, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm